CLINICAL TRIAL: NCT06583694
Title: Bangkok Noi District Electronic Health Database With Socioeconomic Factors From Bangkok Noi Model Project (BANMOP)
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naris Kitnarong, Associate professore, Siriraj Hospital
Other Study IDs: SI002
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Conditions Influencing Health Status; Health Knowledge, Attitudes, Practice; Health-Related Behavior
Keywords: Health Promotion; Elderly; Community health
MeSH Terms: conditions — Behavior; Health Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 0 to 5 year-olds: Participants aged between 0-5 year-olds
  Interventions: Behavioral: Health promotion campaigns to correct the health problems
- 6- 14 year-olds: Participants aged between 6-14 year-olds
  Interventions: Behavioral: Health promotion campaigns to correct the health problems
- 15-21 year-olds: Participants aged between 15-21 year-olds
  Interventions: Behavioral: Health promotion campaigns to correct the health problems
- 22-59 year-olds: Participants aged between 22-59 year-olds.
  Interventions: Behavioral: Health promotion campaigns to correct the health problems
- equal to and more than 60 year-olds: Participants aged equal to and more than 60 year-olds
  Interventions: Behavioral: Health promotion campaigns to correct the health problems

INTERVENTIONS:
Behavioral: Health promotion campaigns to correct the health problems

SUMMARY:
Bangkoknoi Model Project (BANMOP) is guided by context-specific health databases to promote the sustainable health and well-being of people living in the Bangkoknoi district. The BANMOP is a prospective cohort project that emphasizes community engagement via electronic databases. Data were collected from households in Bangkoknoi district. Convenience sampling was used and the data were collected via mobile application and a web-based platform, and by face-to-face interviews with well-trained volunteers who were mainly health professionals. The data were categorized by age groups: 0-5, 6-14, 15-21, 22-59, >60 years old, included both individuals and families in five categories: health, environment & disaster, economics, social, and safety.

DETAILED DESCRIPTION:
A total of 21,286 participants from 42 Bangkoknoi communities accounted for 16.08% of total population of Bangkoknoi district were participated. Forty percent of participants reported having physical health problems. Noncommunicable diseases were dominated by physical health issues as age progressed. Overall, hypertension was the most prevalent health problem at 12.6 % followed by allergic diseases (11%), diabetes mellitus (7.5%), and dyslipidemia (6.1%). Anxiety was the most common mental disorder and gender income disparity is an important issue. Although, 91.6% of participants satisfied with their home environment, but the crowded, cluttered, urban environment caused their dissatisfaction. Forty-two percent reported the problems related to reproductive health such as teen pregnancy (16.72%), family planning and marriage guidance (12.74%), premature sexual transmitted diseases (8.96%) and infertility (3.78%). Subsequently, 17 sub-projects were established to promote the sustainable health and well-being of people in the Bangkoknoi district.

ELIGIBILITY:
The total population of Bangkoknoi district included 132,372 individuals in 48,771 households.

Inclusion Criteria:

1. Individuals registered with the Bangkoknoi district and currently reside there.
2. Individuals who are not registered, but currently reside in the Bangkoknoi district.
3. Individuals registered with the Bangkoknoi district, but who currently reside outside the district.
4. Individuals, both Thai and non-Thai citizens, who work in the Bangkoknoi district continuously for at least 30 days.
5. Individuals who study at schools or universities in the Bangkoknoi district continuously for at least 30 days.

Exclusion Criteria:

* Individuals who were not willing to participate or answer the questionnaires were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The total population of Bangkoknoi district included 132,372 individuals in 48,771 households and (one of the following)
  1. Individuals registered with the Bangkoknoi district and currently reside there.
  2. Individuals who are not registered, but currently reside in the Bangkoknoi district.
  3. Individuals registered with the Bangkoknoi district, but who currently reside outside the district.
  4. Individuals, both Thai and non-Thai citizens, who work in the Bangkoknoi district continuously for at least 30 days.
  5. Individuals who study at schools or universities in the Bangkoknoi district continuously for at least 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 21286 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
health conditions | 4.5 years from 1st of October 2015 to the 31st of March 2020
  survey questionnaires on individual and household health condition

SECONDARY OUTCOMES:
Health-related conditions | 4.5 years from 1st of October 2015 to the 31st of March 2020
  survey questionnaires on individual and household health-related condition including environment & disaster, economics, social, and safety

CONTACTS AND LOCATIONS:
Overall Officials: Naris Kitnarong, M.D., M.B.A., Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: Yes
All IPD could be shared under reasonable request via the website: www.bangkoknoimodel.com
Supporting Information: SAP, CSR
Time Frame: Since March 2020 to up to 10 years after
Access Criteria: For non-profit organizations only. For further projects/researches that related to Bangkoknoi area/individuals
URL: https://www.bangkoknoimodel.com/stat.

REFERENCES:
- [Result] Wiles JL, Leibing A, Guberman N, Reeve J, Allen RE. The meaning of "aging in place" to older people. Gerontologist. 2012 Jun;52(3):357-66. doi: 10.1093/geront/gnr098. Epub 2011 Oct 7. PMID 21983126
- [Result] Atthawuttikul, A., 2016. Comparison of Elderly People's Perception of Homely Feeling towards Room Environment in Their Own Home and in Two Nursing Homes in Thailand. International Journal of Social Science and Humanity, 6(11), pp.865-868.
- [Derived] Kitnarong N, Muangpaisan W, Kaweewongprasert P, Luerithiphong S, Apinuntavech S, Manaboriboon B, Talungchit P, Chainuvati S, Srinonprasert V, Kade S, Supamanee K, Assantachai P, Watanapa P. Electronic health databases and surveys for community-specific health promotion, prevention, and interventions: the Bangkoknoi Model Project (BANMOP). BMC Health Serv Res. 2025 May 10;25(1):678. doi: 10.1186/s12913-025-12837-z. PMID 40349067
- See also: Bangkoknoi model Research protocol and data analysis — https://www.bangkoknoimodel.com/stat.
- Available data/document: Clinical Study Report — https://www.bangkoknoimodel.com/stat.